CLINICAL TRIAL: NCT04640558
Title: The Relationship Between Gluteus Medius Latent Trigger Point and Muscle Strength in Healthy Subjects
Brief Title: Gluteus Medius Latent Trigger Point and Muscle Strength in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Medical Doctor, Kars State Hospital
Other Study IDs: KarsSH
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Myofascial Pain Syndrome; Muscle Weakness
Keywords: Trigger point; Gluteus medius muscle
MeSH Terms: conditions — Myofascial Pain Syndromes; Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1. Latent Myofascial Trigger Point Group: 24 participants who will be clinically diagnosed with unilateral latent myofascial trigger point in the dominant side gluteus medius muscle.
  Interventions: Device: Muscle strength measurement
- Group 2. Non-Latent Myofascial Trigger Point Group: 24 participants who don't have latent myofascial trigger point.
  Interventions: Device: Muscle strength measurement

INTERVENTIONS:
Device: Muscle strength measurement — The bilateral gluteus medius muscle strength of each participant will be measured by the assessor (MB) blinded to the participants using the Lafayette manual muscle tester. (Lafayette Instrument Company, Lafayette IN, USA). In the participant's side-lying position, the practitioner applied resistance from the upper ankle to the abduction movement with slight flexion of the upper hip. During the measurements, the participants were asked to perform the maximum isometric contraction for 3 seconds. Gluteus medius muscle strength measurements were repeated three times, one minute apart, on the right and left sides. The mean of the measurements was calculated and recorded

SUMMARY:
This study aimed to investigate the relationship between latent MTrPs and gluteus medius muscle strength in a group of healthy adults.

DETAILED DESCRIPTION:
Latent myofascial trigger points (MTrPs) do not cause spontaneous pain; however, they may lead to a limited range of motion and muscle weakness. We hypothesized that latent MTrPs might decrease gluteus medius muscle strength in healthy individuals. Forty-eight healthy men will be included in the study. Trigger point examination for the gluteus medius will be performed bilaterally. Subjects with one or more trigger points on the dominant side and those without any trigger points will be assigned to two groups. Muscle strength for gluteus medius will be assessed with a manual muscle tester using the "break test" technique on both sides. The subjects and the examiners will be blinded. For statistical analysis, the independent sample t-test was used to compare the intergroup differences.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: 18-40 years.
* Absence of musculoskeletal complaints related to the lumbar, sacroiliac, and hip area.
* Absence of bilateral latent MTrP in the gluteus medius muscle.
* Latent trigger point in the gluteus medius muscle on the dominant side with palpation.

Exclusion Criteria:

* A history of medical treatment, physical therapy, injection therapy, or surgical treatment related to the lumbar, sacroiliac, and hip area.
* History of trauma, or malignancy or being pregnant, or if the patient is in the lactation period.
* Bilateral latent MTrP in the gluteus medius muscle.
* Presence of latent MTrP on the non-dominant side.

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: 24 participants who are clinically diagnosed with unilateral latent MTrP in the dominant side gluteus medius muscle and 24 participants who don't have latent MTrP.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
Gluteus medius muscle strength | One month
  In the participant's side-lying position, the practitioner will be applied resistance from the upper ankle to the abduction movement with slight flexion of the upper hip. During the measurements, the participants will be asked to perform the maximum isometric contraction for 3 seconds. Gluteus medius muscle strength measurements will be repeated three times, one minute apart, on the right and left sides. The mean of the measurements will be calculated and recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No